CLINICAL TRIAL: NCT01124292
Title: Development and Translational Assessment of a Tongue-Based Assistive Neuro-Technology for Individuals With Severe Neurological Disorders
Brief Title: Evaluation of a Tongue Operated Assistive Technology for Individuals With Severe Paralysis
Acronym: TDS-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Shepherd Center, Atlanta GA (Other); Northwestern University (Other); Shirley Ryan AbilityLab (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Maysam Ghovanloo, Associate Processor, Georgia Institute of Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H09240; 1RC1EB010915-01 (NIH)
Record Dates: First submitted 2010-05-10; First posted 2010-05-17 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Quadriplegia; Spinal Cord Injury; ALS
Keywords: Disability; Quadriplegia; Paralysis; Assistive technology; Quality of life; Computer access; Wheeled mobility
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries; Paralysis | interventions — Body Piercing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Able-bodied subject with piercing (Experimental): Able-bodied subjects who already have tongue piercing.
  Interventions: Device: Usability assessment
- Able-bodied subject without piercing (Experimental): Able-bodied subjects who willing to receive a tongue piercing for this study.
  Interventions: Procedure: Tongue Piercing; Device: Usability assessment
- Subjects with spinal cord injury (Experimental): Persons with mobility limitations requiring power wheel chair, able to move tongue, able to follow simple commands, and have some experience with computers. All participants willingly received a mid-line tongue piercing.
  Interventions: Procedure: Tongue Piercing; Device: Usability assessment

INTERVENTIONS:
Procedure: Tongue Piercing — Subjects brush their teeth, and then swish and spit with chlorhexidine mouthwash for 30-60s. Subjects would be placed in a semirecumbent position in a procedure chair. After marking the piercing site using a sterilized surgical marking pen the protruded tongue would be pierced. Anesthesia may be used during the piercing at the discretion of the operator and the subject. A sterilized titanium or surgical grade stainless steel piercing tongue stud would be placed in an appropriate position on the tongue to minimize complications from the piercing but also facilitate good functionality of the TDS.
  Arms: Able-bodied subject without piercing; Subjects with spinal cord injury
Device: Usability assessment — Computer access: Subjects wear the TDS and get trained. Then they sit 1.5 m from a 22" LCD monitor. Then they use TDS to conduct several tasks using their tongues, such as clicking on target objects and navigating through on-screen maze, while the computer registers their tongue commands and measures their performance.
  Wheelchair control: Subjects wear the TDS and use it to drive an electrically powered wheelchair through an obstacle course using their tongues. The operator measured the time it takes for the subjects to drive through the course as well as the number of collisions.

SUMMARY:
This study was intended to evaluate a new assistive neuro-technology, known as the Tongue Drive System (TDS), by its potential end-users, i.e. individuals with severe disabilities, who are the best experts for indicating the benefits and possible shortcomings of any new ANT. Our goal is to assess the acceptability and usability of the TDS for various tasks that are important in daily lives of these individuals, such as computer access, wheeled mobility, and environmental control.

DETAILED DESCRIPTION:
A new assistive neuro-technology (ANT), called the Tongue Drive System (TDS), enables individuals with severe disability access their environment with nothing but their tongue motion. The human tongue is inherently capable of sophisticated control and manipulation tasks with many degrees of freedom. It can move rapidly and accurately within the mouth such that the tip can touch every single tooth. The direct connection between the brain and the tongue generally allows it to escape damage even in severe spinal cord injuries (SCI). Unlike the brain, the tongue is accessible, and its location inside the mouth affords a degree of privacy.

TDS consists of a magnetic tracer, the size of a lentil, attached to the tongue by gluing, implantation, or piercing. The tracer generates a magnetic field inside and around the mouth that is detected by an array of magnetic sensors mounted on a wireless headset. Tongue-movement-induced changes in the magnetic field are sent wirelessly to an ultra-mobile computer or smartphone, carried by the user, which processes and translates every tongue motion to a particular user-defined function.

Once an individual with disability is "enabled" to access a computing device, he/she can nearly do everything that an able-bodied individual can do with that device. This includes communicating, education, training, entertainment, and controlling other devices such as powered wheelchairs (PWC), assistive robotic manipulators, and other home/office appliances on a local area network (LAN). Even the individual's own natural or prosthetic limbs can be manipulated to move by functional electrical stimulation (FES).

This study was intended to evaluate the TDS by the ultimate intended users, individuals with severe disabilities, who are the best experts for indicating the benefits and possible shortcomings of any new ANT. Our goal is to assess the acceptability and usability of the TDS for various tasks that are important in daily life such as computer access, wheeled mobility, and environmental control.

Three groups of subjects were recruited:

Group-A: Able-bodied subjects who already have tongue piercing

Group-B: Able-bodied subjects who wanted to receive tongue piercing as part of this trial

Group-C: Subjects with high-level disability, who wanted to receive tongue piercing as part of this trial

Each group of subjects participated in a battery of tasks that quantitatively measures their performance in accessing computers and driving wheelchairs using the TDS.

We also devised acceptable procedures for receiving a magnetic tongue piercing (required in order to use the TDS), and assess its potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

Inclusion group-A:

* Age 18-65
* Able-bodied with a tongue piercing Must have had the tongue piercing for at least 3 months and still be using it
* Piercing is located in the midline of the tongue between the tip and the frenulum, almost in the center of the mouth
* Can understand and speak English
* Have some experience in using computers

Inclusion group-B:

* Age 18-65
* No overt sign of disability or neurological disease
* Do not have a tongue piercing, but are willing to receive one in the midline between the tip and lingual frenulum, almost in the center of the mouth
* Can understand and speak English
* Have some experience in using computers

Inclusion group-C:

* Age 18-65
* Have mobility limitations requiring a power wheel chair and also have inadequate upper limb strength to manage a hand or arm control i.e. have severe motor disabilities and need alternative control
* Either using or suitable for an alternative control
* Able to follow simple commands
* Sitting tolerance of at least 4 hours (each experiment session will be no more than 4 hours and the researcher follows the standard pressure relief schedule)
* Have some experience in using computers
* Be able to move the tongue
* Be able to speak or respond to questions by themselves or through an augmentative and alternative communication (AAC) device
* Be able to give consent
* Be able to have a caregiver, who can respond immediately in the event of an emergency, available during the period of the study.
* Can understand and speak English
* Have or are willing to receive a tongue piercing in the midline between the tip and the lingual frenulum, almost in the center of the mouth

Exclusion Criteria:

Exclusion Group-A:

* Original tongue piercing and the insertion site is too wide.
* Ongoing difficulties with current tongue jewelry
* Tongue piercing not located in the correct position on the tongue
* No experience with computers or illiterate
* Severe hearing or visual deficiency or impairing neurological disease
* Have any ongoing systemic condition deemed to be relevant by the local investigator-clinician
* Is pregnant
* Cognitive impairment so that unable to follow simple commands
* Wounds or ulcers on the head or in the mouth or on the tongue
* Using sensitive electronic implantable medical device such as a deep brain stimulator or a pacemaker in the upper body
* Intra-oral space occupying lesion or orthodontic appliance
* Unable to come to GT or RIC on a regular basis during the study-period
* Miss more than two appointments without prior notification
* Unable to comply with any of the procedures in the protocol

Exclusion Group-B:

* Tongue too short or the tongue web too far extended, making tongue piercing difficult
* Have a torus mandibularis or palatini or other space-occupying intra-oral lesion or orthodontic appliance
* No experience with computers or illiterate
* Severe hearing or visual deficiency or impairing neurological disease
* Cardiovascular and respiratory diseases, artificial heart valve, congenital heart disease
* On an immunosuppressive medication or otherwise immunocompromised
* Diabetic or have any other ongoing systemic condition deemed to be relevant by the local investigator-clinician
* Ongoing neoplastic disease other than localized basal cell or squamous cell carcinoma of the skin
* Have known asthma, physical urticaria or angioedema
* Have any current infectious condition
* Cognitive impairment to the extent that cannot follow simple commands
* Is pregnant
* Wounds or ulcers on the head or in the mouth or on the tongue
* Using sensitive electronic implantable medical device such as a deep brain stimulator or a pacemaker in the upper body
* Space occupying orthodontic appliances
* Unable to come SCA or NU for a tongue piercing, 72 hour visit and to GTB or RIC on a regular basis during the study-period
* Miss more than two appointments without prior notification
* Unable to comply with any of the procedures in the protocol

Exclusion Group-C:

* Unable to move the tongue
* Have a large object or tube in the mouth blocking tongue motion
* Tongue or tongue frenulum short or the tongue frenulum extended far forward, making tongue piercing difficult
* Have a torus mandibularis or palatini or other space-occupying intra-oral lesion or orthodontic appliance
* Medically or mentally unstable
* Known sensitivity or allergy to an adhesive
* Using a halo brace or facial pads that would block the use of a headset or headgear
* Cognitive impairment to the extent that the subject cannot follow simple commands
* Severe hearing or visual deficiency
* Cardiovascular and respiratory diseases, artificial heart valve, congenital heart disease
* On any form of anticoagulation including but not limited to warfarin, heparin, low-molecular-weight heparin, factor Xa inhibitors, aspirin, aspirin-containing products, or nonsteroidal anti-inflammatory medications that the subject's supervising attending physician states cannot be stopped during the pre-piercing period which may include not only the appropriate medication-specific washout period before the piercing but also up to 5 days after the procedure.
* On an immunosuppressive or otherwise immunocompromised
* Have a decubitus ulcer stage III or higher or a decubitus ulcer of any stage that is worsening.
* Diabetic or have any other ongoing systemic condition, as deemed to be relevant by the local investigator-clinician
* Ongoing neoplastic disease other than localized basal cell or squamous cell carcinoma of the skin
* Have known asthma, physical urticaria or angioedema
* Have any current infectious condition
* Is pregnant
* No experience with computers or illiterate
* Using a sensitive electronic implantable medical device such as a deep brain stimulator or a pacemaker in the upper body
* Unable to sit for 4 hours with pressure relief
* Wounds or ulcers on the head or in the mouth or on the tongue
* No continuous access to a caregiver
* Unable to come to the SCA or NMH for a three day stay for tongue piercing and to SCA or RIC on a regular basis during the study-period
* Miss more than three appointments without prior notification
* Unable to comply with any of the procedures in the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maysam Ghovanloo, Ph.D., Principal Investigator — Georgia Institute of Technology
Locations (4):
- United States (4):
  - Georgia Institute of Technology, Atlanta, Georgia
  - Shepherd Center, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rehabilitation Institute of Chicago, Chicago, Illinois

REFERENCES:
- [Background] Huo X, Ghovanloo M. Evaluation of a wireless wearable tongue-computer interface by individuals with high-level spinal cord injuries. J Neural Eng. 2010 Apr;7(2):26008. doi: 10.1088/1741-2560/7/2/026008. Epub 2010 Mar 23. PMID 20332552
- [Background] Huo X, Ghovanloo M. Using unconstrained tongue motion as an alternative control mechanism for wheeled mobility. IEEE Trans Biomed Eng. 2009 Jun;56(6):1719-26. doi: 10.1109/TBME.2009.2018632. Epub 2009 Apr 7. PMID 19362901
- [Background] Huo X, Wang J, Ghovanloo M. Introduction and preliminary evaluation of the Tongue Drive System: wireless tongue-operated assistive technology for people with little or no upper-limb function. J Rehabil Res Dev. 2008;45(6):921-30. doi: 10.1682/jrrd.2007.06.0096. PMID 19009478
- [Background] Huo X, Wang J, Ghovanloo M. A magneto-inductive sensor based wireless tongue-computer interface. IEEE Trans Neural Syst Rehabil Eng. 2008 Oct;16(5):497-504. doi: 10.1109/TNSRE.2008.2003375. PMID 18990653
- [Background] Huo X, Ghovanloo M. Using speech recognition to enhance the Tongue Drive System functionality in computer access. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:6393-6. doi: 10.1109/IEMBS.2011.6091578. PMID 22255801
- [Result] Yousefi B, Huo X, Veledar E, Ghovanloo M. Quantitative and comparative assessment of learning in a tongue-operated computer input device. IEEE Trans Inf Technol Biomed. 2011 Sep;15(5):747-57. doi: 10.1109/TITB.2011.2158608. Epub 2011 Jun 7. PMID 21652288
- [Result] Yousefi B, Huo X, Kim J, Veledar E, Ghovanloo M. Quantitative and comparative assessment of learning in a tongue-operated computer input device--part II: navigation tasks. IEEE Trans Inf Technol Biomed. 2012 Jul;16(4):633-43. doi: 10.1109/TITB.2012.2191793. Epub 2012 Jun 6. PMID 22692932
- [Result] Kim J, Huo X, Minocha J, Holbrook J, Laumann A, Ghovanloo M. Evaluation of a smartphone platform as a wireless interface between tongue drive system and electric-powered wheelchairs. IEEE Trans Biomed Eng. 2012 Jun;59(6):1787-96. doi: 10.1109/TBME.2012.2194713. Epub 2012 Apr 16. PMID 22531737
- [Derived] Minocha JS, Holbrook JS, West DP, Ghovanloo M, Laumann AE. Development of a tongue-piercing method for use with assistive technology. JAMA Dermatol. 2014 Apr;150(4):453-4. doi: 10.1001/jamadermatol.2013.7165. No abstract available. PMID 24284925
- See also: CNN report on the first clinical trial of the Tongue Drive System at the Shepherd Center in 2009 — http://www.cnn.com/2010/HEALTH/01/25/hm.wheelchair.tongue/index.html
- See also: Tongue Drive System featured on the Science Nation (the National Science Foundation online Magazine), showing a short video clip of the first clinical trial at the Shepherd Center in Atlanta. — http://www.nsf.gov/news/special_reports/science_nation/tonguedriver.jsp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Able-bodied subjects (groups A and B) were recruited by using local IRB-approved flyers, emails, and electronically distributed documents.
  Subjects with spinal cord injuries were recruited from the in- and outpatient departments of the Shepherd Center and the Rehabilitation Institute of Chicago.
  (May. 2010 - March. 2012)
Groups:
- Able-bodied Subject With Tongue Piercing: Able-bodied subjects who already have tongue piercing.
- Able-bodied Subject Without Tongue Piercing: Able-bodied subjects who willing to receive a tongue piercing for this study.
Period: Overall Study
Arm/Group | Able-bodied Subject With Tongue Piercing | Able-bodied Subject Without Tongue Piercing | Subjects With Spinal Cord Injury
Started | 16 | 24 | 21
Completed | 14 | 9 | 11
Not Completed | 2 | 15 | 10
Not completed — Lost to Follow-up | 2 | 4 | 3
Not completed — Physician Decision | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 6 | 2
Not completed — medical issue unrelated to the study | 0 | 0 | 2
Not completed — piercing track closed | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Able-bodied Subject Without Tongue Piercing:: Able-bodied subjects who willing to receive a tongue piercing for this study.
- Total: Total of all reporting groups
Arm/Group | Able-bodied Subject With Tongue Piercing | Able-bodied Subject Without Tongue Piercing: | Subjects With Spinal Cord Injury | Total
Number analyzed (Participants) | 14 | 9 | 11 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 13 | 9 | 11 | 33
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.12 (4.85) | 22.56 (4.00) | 38.30 (10.25) | 27.61 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 2 | 17
  Male | 4 | 4 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 9 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Fitts' Law: Horizontal Tapping Using TDS, Keypad, and Mouse (Throughput)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Horizontal Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. This data was then fed into an equation, which provided the throughput measure. The unit of throughput is "bits per second".
  The high value of throughput means better performance. Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: bits per second
Groups:
- Able-bodied Subject With Tongue Piercing (Group-A): Able-bodied subjects who already have tongue piercing.
- Able-bodied Subject Without Tongue Piercing (Group-B): Able-bodied subjects who willing to receive a tongue piercing for this study.
- Subjects With Spinal Cord Injury (Group-C): Persons with mobility limitations requiring power wheel chair, able to move tongue, able to follow simple commands, and have some experience with computers. All participants willingly received a mid-line tongue piercing.
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
bits per second
  first session using TDS | 1.97 (0.44) | 2.03 (0.44) | 1.54 (0.56)
  second session using TDS | 2.04 (0.39) | 2.22 (0.52) | 1.75 (0.42)
  third session using TDS | 2.34 (0.32) | 2.48 (0.51) | 1.90 (0.51)
  fourth session using TDS | 2.37 (0.50) | 2.54 (0.48) | 2.14 (0.54)
  fifth session using TDS | 2.44 (0.52) | 2.47 (0.54) | 2.09 (0.41)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 2.22 (0.51)
  first session using keypad | 2.85 (0.41) | 3.49 (0.68) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 2.96 (0.45) | 3.69 (0.48) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 3.09 (0.52) | 3.84 (0.54) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 3.14 (0.48) | 3.81 (0.59) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 3.17 (0.52) | 3.84 (0.57) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using mouse | 3.89 (0.97) | 4.17 (0.68) | NA (NA) — Subjects with Spinal cord injury cannot use the mouse.

2. Primary Outcome: Fitts' Law: Horizontal Tapping Using TDS, Keypad, and Mouse (Error Rate)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Horizontal Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. The error rate is the rate of outside of targets vs. total targets.
  Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Percentage of Missed Targets (%)
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
Percentage of Missed Targets (%)
  first session using TDS | 29.14 (13.96) | 23.85 (11.04) | 37.84 (21.65)
  second session using TDS | 24.08 (17.30) | 18.36 (10.11) | 30.62 (18.02)
  third session using TDS | 24.64 (14.89) | 13.70 (8.14) | 28.77 (17.72)
  fourth session using TDS | 20.74 (14.36) | 14.90 (9.34) | 24.01 (14.16)
  fifth session using TDS | 17.96 (10.41) | 16.34 (10.26) | 18.45 (9.83)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 19.81 (12.63)
  first session using keypad | 9.49 (7.96) | 10.63 (8.35) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 6.94 (6.21) | 8.44 (7.40) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 6.70 (6.12) | 5.97 (3.96) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 5.03 (4.41) | 8.12 (6.54) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 4.99 (4.27) | 6.24 (5.19) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using mouse | 9.24 (11.91) | 2.14 (2.14) | NA (NA) — Subjects with Spinal cord injury cannot use the mouse.

3. Primary Outcome: Fitts' Law: Vertical Tapping Using TDS, Keypad, and Mouse (Throughput)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Vertical Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. This data was then fed into an equation, which provided the throughput measure. The unit of throughput is "bits per second".
  The high value of throughput means better performance. Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: bits per second
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
bits per second
  first session using TDS | 2.14 (0.41) | 2.22 (0.54) | 1.44 (0.50)
  second session using TDS | 2.27 (0.37) | 2.54 (0.51) | 1.77 (0.54)
  third session using TDS | 2.31 (0.45) | 2.74 (0.30) | 1.79 (0.56)
  fourth session using TDS | 2.44 (0.36) | 2.76 (0.45) | 1.97 (0.33)
  fifth session using TDS | 2.61 (0.30) | 2.69 (0.49) | 2.01 (0.43)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 2.18 (0.60)
  first session using keypad | 2.84 (0.44) | 3.46 (0.61) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 2.90 (0.56) | 3.88 (0.58) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 3.03 (0.45) | 3.85 (0.58) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 3.10 (0.46) | 3.96 (0.65) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 3.11 (0.54) | 3.93 (0.41) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using mouse | 4.28 (0.71) | 4.32 (0.63) | NA (NA) — Subjects with Spinal cord injury cannot use the mouse.

4. Primary Outcome: Fitts' Law: Vertical Tapping Using TDS, Keypad, and Mouse (Error Rate)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Vertical Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. The error rate is the rate of outside of targets vs. total targets.
  Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Percentage of Missed Targets (%)
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
Percentage of Missed Targets (%)
  first session using TDS | 26.16 (15.39) | 19.47 (9.95) | 38.95 (19.61)
  second session using TDS | 21.83 (13.78) | 15.88 (11.74) | 30.37 (17.31)
  third session using TDS | 22.72 (12.43) | 12.67 (7.52) | 26.67 (15.57)
  fourth session using TDS | 20.30 (13.55) | 10.97 (10.06) | 23.77 (11.32)
  fifth session using TDS | 14.77 (11.79) | 10.97 (7.71) | 21.90 (11.35)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 19.99 (12.44)
  first session using keypad | 9.91 (8.92) | 10.43 (7.80) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 8.95 (7.91) | 8.26 (5.72) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 6.16 (6.02) | 6.41 (5.55) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 5.47 (5.42) | 6.00 (4.82) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 5.83 (5.44) | 7.27 (6.01) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using mouse | 5.02 (7.37) | 2.13 (2.28) | NA (NA) — Subjects with Spinal cord injury cannot use the mouse.

5. Primary Outcome: Fitts' Law: Center-Out Tapping Using TDS, Keypad, Mouse, and SnP (Throughput)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Center-out Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. This data was then fed into an equation, which provided the throughput measure. The unit of throughput is "bits per second".
  The high value of throughput means better performance. This task is tested by the TDS, keypad, mouse and the sip-and-puff device (SnP).
  Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: bits per second
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
bits per second
  first session using TDS | 0.83 (0.32) | 0.77 (0.48) | 0.37 (0.21)
  second session using TDS | 1.23 (0.36) | 0.96 (0.49) | 0.52 (0.27)
  third session using TDS | 1.39 (0.26) | 1.10 (0.40) | 0.51 (0.31)
  fourth session using TDS | 1.41 (0.37) | 1.29 (0.50) | 0.73 (0.45)
  fifth session using TDS | 1.58 (0.25) | 1.41 (0.53) | 0.75 (0.45)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 0.81 (0.40)
  first session using keypad | 1.44 (0.46) | 2.13 (0.57) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 1.74 (0.47) | 2.60 (0.44) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 1.82 (0.29) | 2.83 (0.36) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 1.93 (0.32) | 3.02 (0.30) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 2.03 (0.27) | 3.05 (0.53) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using mouse | 3.86 (0.54) | 3.31 (0.50) | NA (NA) — Subjects with Spinal cord injury cannot use the mouse.
  first session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 0.31 (0.20)
  second session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 0.42 (0.20)
  third session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 0.45 (0.19)
  fourth session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 0.51 (0.16)
  fifth session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 0.52 (0.17)
  sixth session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 0.52 (0.19)

6. Primary Outcome: Fitts' Law: Center-Out Tapping Using TDS, Keypad, Mouse, and SnP (Error Rate)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Center-out Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. The error rate is the rate of outside of targets vs. total targets. This task is tested by the TDS, keypad, mouse and the sip-and-puff device (SnP).
  Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Percentage of Missed Targets (%)
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
Percentage of Missed Targets (%)
  first session using TDS | 37.65 (15.14) | 41.41 (20.38) | 61.98 (26.32)
  second session using TDS | 27.33 (12.18) | 32.61 (12.51) | 55.05 (24.75)
  third session using TDS | 23.02 (10.47) | 23.87 (10.39) | 48.15 (25.29)
  fourth session using TDS | 19.71 (10.80) | 25.17 (13.93) | 41.44 (23.40)
  fifth session using TDS | 17.52 (9.15) | 19.84 (8.80) | 36.54 (22.34)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 39.00 (27.32)
  first session using keypad | 12.66 (7.67) | 6.68 (6.38) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 11.81 (8.95) | 4.86 (6.04) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 9.67 (7.61) | 1.33 (1.51) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 7.69 (5.36) | 2.08 (2.57) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 6.72 (4.67) | 2.38 (2.40) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using mouse | 4.46 (5.63) | 2.95 (3.00) | NA (NA) — Subjects with Spinal cord injury cannot use the mouse.
  first session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 42.50 (25.34)
  second session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 31.71 (20.80)
  third session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 26.67 (19.96)
  fourth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 20.69 (15.41)
  fifth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 19.83 (18.00)
  sixth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 16.52 (12.52)

7. Primary Outcome: Fitts' Law: Center-Out Tapping Using TDS, Keypad, Mouse, and SnP (Movement Time)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Center-out Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. The movement time is the cursor movement time from the initial movement to the final movement for each target. This task is tested by the TDS, keypad, mouse and the sip-and-puff device (SnP).
  Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
seconds
  first session using TDS | 1.70 (0.30) | 1.29 (0.15) | 4.00 (1.41)
  second session using TDS | 1.33 (0.17) | 1.22 (0.13) | 3.18 (1.44)
  third session using TDS | 1.30 (0.17) | 1.21 (0.11) | 3.12 (1.38)
  fourth session using TDS | 1.34 (0.24) | 1.22 (0.15) | 2.81 (1.21)
  fifth session using TDS | 1.26 (0.16) | 1.18 (0.08) | 2.75 (1.25)
  sixth session using TDS | NA (NA) — Group-A subjects completed 5-session trials. | NA (NA) — Group-B subjects completed 5-session trials. | 2.75 (1.24)
  first session using keypad | 1.29 (0.15) | 1.29 (0.39) | NA (NA) — Group-C subjects could not use a keypad.
  second session using keypad | 1.22 (0.13) | 0.97 (0.12) | NA (NA) — Group-C subjects could not use a keypad.
  third session using keypad | 1.21 (0.11) | 0.95 (0.14) | NA (NA) — Group-C subjects could not use a keypad.
  fourth session using keypad | 1.22 (0.15) | 0.88 (0.11) | NA (NA) — Group-C subjects could not use a keypad.
  fifth session using keypad | 1.18 (0.08) | 0.87 (0.12) | NA (NA) — Group-C subjects could not use a keypad.
  first session using mouse | 0.66 (0.08) | 0.78 (0.07) | NA (NA) — Group-C subjects could not use a mouse.
  first session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 4.48 (1.08)
  second session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 4.14 (0.90)
  third session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 3.81 (0.71)
  fourth session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 3.69 (0.76)
  fifth session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 3.64 (0.83)
  sixth session using SnP | NA (NA) — Group-A subjects did not test using SnP. | NA (NA) — Group-B subjects did not test using SnP. | 3.79 (0.89)

8. Primary Outcome: Fitts' Law: Multi-Directional Tapping Using TDS, Keypad, and Mouse (Throughput)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Multi-directional Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. This data was then fed into an equation, which provided the throughput measure. The unit of throughput is "bits per second".
  The high value of throughput means better performance. Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: bits per second
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
bits per second
  first session using TDS | 0.40 (0.19) | 0.80 (0.30) | 0.39 (0.17)
  second session using TDS | 0.62 (0.21) | 0.93 (0.31) | 0.42 (0.21)
  third session using TDS | 0.77 (0.30) | 1.05 (0.30) | 0.45 (0.16)
  fourth session using TDS | 0.85 (0.32) | 1.10 (0.26) | 0.65 (0.21)
  fifth session using TDS | 0.98 (0.26) | 1.16 (0.31) | 0.64 (0.27)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 0.73 (0.31)
  first session using keypad | 0.88 (0.28) | 1.44 (0.20) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 1.03 (0.24) | 1.69 (0.20) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 1.11 (0.21) | 1.85 (0.17) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 1.19 (0.18) | 1.86 (0.22) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 1.16 (0.22) | 1.87 (0.23) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using mouse | 4.32 (0.59) | 4.06 (0.60) | NA (NA) — Subjects with Spinal cord injury cannot use the mouse.

9. Primary Outcome: Fitts' Law: Multi-Directional Tapping Using TDS, Keypad, and Mouse (Error Rate)
Description: Subjects used the tongue drive system (TDS) to move the mouse cursor towards targets with various sizes and distances on the computer screen (Multi-directional Tapping task) and select those targets. The computer measured the time it took for the subjects to reach the targets and the accuracy of their selections from the center of the targets. The error rate is the rate of outside of targets vs. total targets.
  Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Percentage of Missed Targets (%)
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
Percentage of Missed Targets (%)
  first session using TDS | 32.67 (19.60) | 21.34 (14.17) | 54.91 (22.34)
  second session using TDS | 21.56 (13.87) | 14.27 (9.69) | 51.52 (27.88)
  third session using TDS | 18.42 (14.28) | 10.73 (8.48) | 37.27 (19.88)
  fourth session using TDS | 18.00 (15.27) | 8.08 (6.67) | 27.88 (25.15)
  fifth session using TDS | 14.67 (13.99) | 6.86 (5.52) | 29.47 (20.13)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 29.10 (24.28)
  first session using keypad | 7.25 (7.36) | 2.62 (3.38) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 6.38 (8.73) | 1.64 (2.36) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 3.99 (6.26) | 1.30 (2.46) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 3.65 (4.77) | 1.84 (2.37) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 4.96 (6.36) | 1.44 (2.06) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using mouse | 6.77 (7.13) | 2.78 (3.21) | NA (NA) — Subjects with Spinal cord injury cannot use the mouse.

10. Primary Outcome: Information Transfer Rate (ITR)
Description: Computer randomly highlights one out of six or four commands and the subjects issue that particular command using the tongue drive system (TDS) and the sip-and-puff device (SnP). Subjects are given a time period (T). The time intervals for the TDS:(Group-A)2.0s,1.5s,1.0s,(Group-B &-C)1.0s,0.7s,0.5s, SnP:(Group-C)1.2s,1.0s,0.7s. The saturated results were observed from the second session during Group-A trials. Therefore, we reduced the time period from the Group-B trial. Moreover, the SnP device needs a certain time period to issue a command and we observed that the minimum possible time period was 0.7 seconds. At the end the percentage of correctly selected commands is calculated and fed into an equation along with the time given to the subjects for each selection.Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: bits per minute
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
bits per minute
  1st ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 74.33 (5.99) | 128.40 (23.44) | 66.68 (25.01)
  2nd ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 75.53 (5.18) | 146.34 (12.40) | 99.15 (41.14)
  3rd ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 74.74 (6.38) | 146.99 (15.44) | 93.62 (32.01)
  4th ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 74.89 (7.04) | 146.29 (14.18) | 112.85 (42.17)
  5th ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 75.47 (6.66) | 146.45 (12.83) | 133.28 (24.46)
  6th ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 127.83 (28.02)
  1st ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 96.13 (14.07) | 184.28 (37.04) | 106.73 (36.05)
  2nd ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 98.29 (8.90) | 208.64 (19.28) | 126.94 (59.05)
  3rd ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 98.14 (10.16) | 208.15 (19.35) | 120.41 (43.85)
  4th ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 100.34 (7.82) | 209.85 (18.94) | 141.27 (53.89)
  5th ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 101.40 (5.50) | 208.45 (20.40) | 164.80 (51.32)
  6th ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 169.31 (51.77)
  1st ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 131.77 (24.28) | 258.08 (47.10) | 114.78 (45.40)
  2nd ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 140.31 (19.85) | 279.59 (39.96) | 141.03 (43.06)
  3rd ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 138.62 (17.13) | 277.63 (42.97) | 110.20 (67.33)
  4th ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 146.82 (16.34) | 282.89 (33.87) | 127.45 (55.50)
  5th ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 146.37 (14.43) | 283.06 (37.54) | 198.45 (77.99)
  6th ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 175.21 (81.23)
  1st ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 24.14 (23.30)
  2nd ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 28.81 (24.00)
  3rd ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 37.34 (21.91)
  4th ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 52.04 (24.45)
  5th ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 54.44 (16.57)
  6th ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 54.70 (23.15)
  1st ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 18.12 (21.88)
  2nd ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 39.87 (31.31)
  3rd ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 52.03 (29.57)
  4th ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 57.79 (22.72)
  5th ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 57.73 (24.68)
  6th ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 55.23 (25.69)
  1st ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 28.81 (35.64)
  2nd ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 40.72 (35.24)
  3rd ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 39.89 (37.63)
  4th ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 54.66 (44.31)
  5th ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 54.30 (30.86)
  6th ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 65.00 (50.28)

11. Primary Outcome: Information Transfer Rate (Percentage of Correctly Completed Commands)
Description: Computer randomly highlights one out of six or four commands and the subjects issue that particular command using the tongue drive system (TDS) and the sip-and-puff device (SnP). Subjects are given a time period (T). The time intervals for the TDS:(Group-A)2.0s,1.5s,1.0s,(Group-B &-C)1.0s,0.7s,0.5s,SnP:(Group-C)1.2s,1.0s,0.7s. The saturated results were observed from the second session during Group-A trials. Therefore, we reduced the time period from the Group-B trial. Moreover, the SnP device needs a certain time period to issue a command and we observed that the minimum possible time period was 0.7 seconds. At the end the percentage of correctly selected commands is calculated and fed into an equation along with the time given to the subjects for each selection.Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Percentage of correctly completed cmd(%)
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
Percentage of correctly completed cmd(%)
  1st ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 98.62 (2.61) | 93.51 (1.24) | 73.87 (11.72)
  2nd ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 99.12 (2.30) | 98.15 (0.51) | 83.70 (15.37)
  3rd ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 98.75 (3.03) | 98.73 (0.45) | 83.93 (9.60)
  4th ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 98.75 (3.45) | 98.08 (0.61) | 90.95 (10.80)
  5th ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | 99.79 (1.58) | 98.17 (0.54) | 94.63 (6.60)
  6th ses. using TDS (Grp A:T=2.0s, Grp B&C T=1.0s) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 93.00 (7.64)
  1st ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 97.50 (5.46) | 93.18 (1.25) | 96.92 (8.85)
  2nd ses. using TDS (Grp A:T=1.5, Grp B&C T=0.7s) | 98.33 (2.99) | 98.06 (0.57) | 82.54 (14.00)
  3rd ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 98.20 (3.65) | 97.99 (0.57) | 78.70 (11.02)
  4th ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 98.97 (2.69) | 98.24 (0.56) | 85.00 (11.75)
  5th ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | 99.37 (1.73) | 98.01 (0.63) | 91.47 (7.93)
  6th ses. using TDS (Grp A:T=1.5s, Grp B&C T=0.7s) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 89.71 (11.71)
  1st ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 94.61 (6.69) | 93.67 (1.25) | 69.34 (12.83)
  2nd ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 96.53 (4.94) | 96.44 (0.99) | 73.91 (8.11)
  3rd ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 94.32 (3.99) | 96.12 (1.05) | 67.66 (16.01)
  4th ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 98.07 (4.04) | 96.96 (0.77) | 72.99 (13.34)
  5th ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | 98.07 (3.28) | 96.87 (0.89) | 84.87 (11.87)
  6th ses. using TDS (Grp A:T=1.0s, Grp B&C T=0.5s) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 78.81 (14.70)
  1st ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 56.48 (22.92)
  2nd ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 62.65 (19.53)
  3rd ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 73.51 (15.05)
  4th ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 79.72 (13.96)
  5th ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 82.41 (9.05)
  6th ses. using SnP (Grp C T=1.2s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 82.72 (10.57)
  1st ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 56.48 (21.85)
  2nd ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 62.65 (25.88)
  3rd ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 75.89 (15.44)
  4th ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 80.00 (12.11)
  5th ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 78.40 (11.15)
  6th ses. using SnP (Grp C T=1.0s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 73.81 (16.62)
  1st ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 43.21 (26.15)
  2nd ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 54.63 (26.49)
  3rd ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 52.78 (24.40)
  4th ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 63.06 (28.17)
  5th ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 62.96 (21.72)
  6th ses. using SnP (Grp C T=0.7s) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 62.78 (26.15)

12. Primary Outcome: On-screen Maze Using TDS, Keypad, and SnP (Completion Time)
Description: Subjects were instructed to use four directional commands (Left, Right, Up, and Down) to move the mouse cursor using the tongue drive system (TDS), keypad, and the sip-and-puff device (SnP) as fast and accurately as possible on a maze. One out of eight maze patterns was randomly selected in each round. The performance measures were completion time (CT) from start to end and sum of deviation (SoD) from the track. SoD was calculated as the sum of all areas between the actual trajectory of the cursor when it was out of the track and the closest edge of the track divided by 1000.
  Group-A and -B were scheduled for five consecutive TDS trials with intervals ranging from two to ten days. Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
seconds
  first session using TDS | 27.80 (18.77) | 23.36 (9.87) | 34.27 (13.25)
  second session using TDS | 16.61 (4.35) | 17.13 (5.72) | 28.71 (12.58)
  third session using TDS | 15.41 (3.45) | 16.81 (12.28) | 32.70 (21.24)
  fourth session using TDS | 15.04 (3.57) | 13.03 (4.49) | 25.93 (9.91)
  fifth session using TDS | 14.26 (2.77) | 12.59 (3.41) | 25.99 (15.27)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 19.47 (14.66)
  first session using keypad | 20.26 (4.21) | 17.56 (6.24) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 16.76 (3.30) | 13.14 (2.34) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 15.30 (2.54) | 12.31 (2.08) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 14.65 (1.67) | 11.76 (2.12) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 14.25 (1.42) | 10.96 (1.99) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 49.86 (28.22)
  second session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 37.48 (18.15)
  third session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 33.49 (12.42)
  fourth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 30.56 (10.08)
  fifth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 30.65 (9.28)
  sixth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 30.89 (10.33)

13. Primary Outcome: On-screen Maze Using TDS, Keypad, and SnP (Sum of Deviation / 1000)
Description: as for outcome 12
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: pixel^2/1000
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
pixel^2/1000
  first session using TDS | 30.05 (89.76) | 23.59 (20.28) | 64.86 (91.42)
  second session using TDS | 4.51 (4.08) | 13.27 (20.28) | 41.86 (41.83)
  third session using TDS | 4.17 (5.20) | 13.91 (31.22) | 59.19 (84.68)
  fourth session using TDS | 4.54 (5.18) | 5.89 (13.05) | 28.43 (24.97)
  fifth session using TDS | 1.80 (1.68) | 4.27 (3.58) | 29.05 (35.49)
  sixth session using TDS | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 17.18 (29.84)
  first session using keypad | 1.88 (2.32) | 4.03 (5.85) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  second session using keypad | 1.10 (1.48) | 1.46 (1.82) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  third session using keypad | 0.60 (1.01) | 1.08 (1.01) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fourth session using keypad | 0.56 (0.66) | 1.55 (1.40) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  fifth session using keypad | 0.39 (0.60) | 1.16 (1.57) | NA (NA) — Subjects with Spinal cord injury cannot use the keypad.
  first session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 47.05 (104.05)
  second session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 20.26 (18.68)
  third session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 14.04 (11.87)
  fourth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 12.19 (11.27)
  fifth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 15.32 (19.02)
  sixth session using SnP | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 11.17 (9.06)

14. Primary Outcome: Driving a Wheelchair Using TDS vs SnP (Completion Time)
Description: An obstacle course will be laid out in an open space and the subjects drive an electric powered wheelchair using the tongue drive system (TDS) and the sip-and-puff device (SnP) to drive through the obstacle course. The operator measured the amount of time it takes for the subjects to begin and return back to the starting point and counts the number of collisions with the obstacles.
  Unlatched and latched: utilize four TDS commands for forward, backward, left, and right motions.
  Unlatched: hold their tongue to keep the PWC moving. Latched: (5 linear speed levels:Backward, Stop, Forward-1, Forward-2, and Forward-3) Issuing the forward or backward commands can increase or decrease the linear speed.
  Semi-proportional: Quickly touching the left and right cheeks- forward or backward commands, sliding tongue over the lip- steer the PWC to the left or right.
  Group-A&-B:5 consecutive TDS trials (intervals ranging from two to ten days) Group-C:computer and PWC within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
seconds
  first session using TDS (unlatched) | 198.17 (34.01) | 240.85 (81.77) | 253.45 (70.11)
  second session using TDS (unlatched) | 169.21 (25.08) | 194.93 (29.48) | 219.46 (56.02)
  third session using TDS (unlatched) | 173.46 (30.27) | 179.39 (29.80) | 186.04 (18.25)
  fourth session using TDS (unlatched) | 170.00 (38.80) | 179.74 (22.78) | 183.70 (23.27)
  fifth session using TDS (unlatched) | 160.08 (18.22) | 154.59 (23.52) | 181.24 (27.39)
  sixth session using TDS (unlatched) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 170.76 (19.76)
  first session using TDS (latched) | 230.29 (48.45) | 260.86 (84.97) | 295.54 (151.08)
  second session using TDS (latched) | 192.46 (27.50) | 210.22 (34.42) | 264.78 (107.65)
  third session using TDS (latched) | 196.08 (35.78) | 200.96 (39.60) | 228.78 (101.65)
  fourth session using TDS (latched) | 181.42 (26.28) | 193.75 (37.92) | 217.63 (84.98)
  fifth session using TDS (latched) | 179.13 (23.22) | 174.33 (34.15) | 189.52 (19.68)
  sixth session using TDS (latched) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 179.37 (23.16)
  first session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 234.97 (70.94)
  second session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 213.28 (68.29)
  third session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 196.24 (37.78)
  fourth session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 183.98 (36.22)
  fifth session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 191.43 (38.12)
  sixth session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 182.33 (21.34)
  first session using TDS (semi-pro) | 196.54 (16.46) | 232.75 (66.47) | 319.21 (112.70)
  second session using TDS (semi-pro) | 178.58 (14.42) | 205.44 (32.64) | 239.18 (62.38)
  third session using TDS (semi-pro) | 177.75 (11.87) | 206.71 (30.35) | 233.92 (60.00)
  fourth session using TDS (semi-pro) | 178.83 (14.70) | 196.57 (28.86) | 212.67 (44.90)
  fifth session using TDS (semi-pro) | 175.25 (17.07) | 177.50 (37.44) | 181.18 (27.27)
  sixth session using TDS (semi-pro) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 204.96 (35.23)

15. Primary Outcome: Driving a Wheelchair Using TDS vs SnP (Number of Navigation Errors)
Description: as for outcome 14
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: Navigation Errors
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 14 | 9 | 11
Navigation Errors
  first session using TDS (unlatched) | 2.67 (1.87) | 8.44 (5.78) | 8.76 (5.04)
  second session using TDS (unlatched) | 1.17 (1.30) | 6.59 (6.76) | 7.48 (4.85)
  third session using TDS (unlatched) | 1.08 (0.79) | 3.96 (4.07) | 5.82 (5.04)
  fourth session using TDS (unlatched) | 1.04 (1.46) | 2.58 (2.26) | 5.06 (4.03)
  fifth session using TDS (unlatched) | 0.75 (0.66) | 2.22 (2.14) | 2.97 (3.56)
  sixth session using TDS (unlatched) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 2.76 (3.46)
  first session using TDS (latched) | 3.50 (2.06) | 7.80 (6.41) | 10.61 (7.61)
  second session using TDS (latched) | 1.83 (1.13) | 6.00 (2.77) | 7.16 (5.00)
  third session using TDS (latched) | 1.38 (1.17) | 4.79 (2.72) | 7.03 (7.26)
  fourth session using TDS (latched) | 0.71 (1.06) | 3.71 (3.16) | 6.78 (9.51)
  fifth session using TDS (latched) | 0.96 (1.44) | 3.70 (3.60) | 3.06 (3.17)
  sixth session using TDS (latched) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 2.06 (2.26)
  first session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 4.27 (3.06)
  second session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 3.30 (2.01)
  third session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 3.82 (2.92)
  fourth session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 2.39 (2.59)
  fifth session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 2.97 (2.30)
  sixth session using SnP (latched) | NA (NA) — Group-A subjects did not test using the SnP. | NA (NA) — Group-B subjects did not test using the SnP. | 2.61 (2.16)
  first session using TDS (semi-pro) | 2.08 (1.23) | 2.52 (1.41) | 7.81 (3.94)
  second session using TDS (semi-pro) | 1.00 (0.91) | 2.92 (1.76) | 5.79 (3.85)
  third session using TDS (semi-pro) | 0.96 (0.84) | 2.00 (2.52) | 5.15 (3.76)
  fourth session using TDS (semi-pro) | 1.00 (1.18) | 1.89 (0.96) | 3.64 (2.97)
  fifth session using TDS (semi-pro) | 0.88 (1.04) | 1.71 (1.69) | 2.97 (3.56)
  sixth session using TDS (semi-pro) | NA (NA) — Group-A subjects completed five-session trials. | NA (NA) — Group-B subjects completed five-session trials. | 3.12 (3.20)

16. Primary Outcome: Phone Dialing Using the Tongue Drive System (TDS) for People With Spinal Cord Injuries (Completion Time)
Description: Randomly selected ten-digit target phone number was visually prompted on the top of the smartphone screen, and the subject entered the same number in the following line as quickly and as accurately as possible. If the wrong number was registered, then the subjects were allowed to delete the one by issuing the deleting command.At the end of the number entering, the subject needs to move the cursor at the green colored "CALL" button, in the middle of the bottom line, and it should be selected to complete the trial. The completion time and error rate were considered to evaluate the performance.
  Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 11
seconds
  first session using TDS | 187.69 (66.09)
  second session using TDS | 109.11 (47.05)
  third session using TDS | 89.99 (21.08)
  fourth session using TDS | 88.37 (29.56)
  fifth session using TDS | 89.37 (27.05)
  sixth session using TDS | 81.87 (22.75)

17. Primary Outcome: Weight Shifting Using the Tongue Drive System (TDS) for People With Spinal Cord Injuries (Completion Time)
Description: The TDS commands were designated to change the wheelchair mode from driving to tilting and to control the wheelchair angle. The completion time was from the initial mode change to the end of the weight shifting.
  Testing sessions for Group-C were divided into computer access and PWC navigation within a week, over 6 weeks.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Subjects With Spinal Cord Injury (Group-C)
Number analyzed (Participants) | 11
seconds
  first session using TDS | 116.19 (42.69)
  second session using TDS | 74.82 (39.10)
  third session using TDS | 78.24 (29.93)
  fourth session using TDS | 75.52 (29.60)
  fifth session using TDS | 74.46 (32.67)
  sixth session using TDS | 71.35 (23.22)

18. Primary Outcome: Short Questionnaire at the End of Each Session Group-A&-B:5 Consecutive TDS Trials (Intervals Ranging From Two to Ten Days) Group-C:Computer and PWC Within a Week, Over 6 Weeks.
Description: Q1.How much thought was necessary to decide where to put your tongue to issue a specific command?1:A lot,5:A Little Q2.Was the speed of the movement of the cursor on the computer screen:1:Too slow,3:Just right,5:Too fast Q3.How difficult was pointing accurately at specific targets on the computer screen?1:Very difficult,5:Very easy Q4.Accurately guiding the powered wheelchair through the obstacle course was:1:Very difficult,5:Very easy Q4.Accurately guiding the powered wheelchair through the obstacle course was:1: Very difficult,5:Very easy (TDS:Q4-1.Unlatched,Q4-2.Latched,Q4-3.Semi-pro,SnP:Q4-4.Latched) Q5.Was the speed of the wheelchair:1:Too slow,5:Too fast Q6.Was the movement of the wheelchair:1:Very jerky,5:Very smooth Q7.Was TDS effective in dialing phone numbers:1:Completely ineffective,5:Very effective Q8.Was TDS effective in doing the weight shift:1:Completely ineffective,5:Very effective
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Subjects With Spinal Cord Injury (Group-C): Computer Session; Subjects With Spinal Cord Injury (Group-C): Wheelchair Session: Persons with mobility limitations requiring power wheel chair, able to move tongue, able to follow simple commands, and have some experience with computers. All participants willingly received a mid-line tongue piercing.
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C): Computer Session | Subjects With Spinal Cord Injury (Group-C): Wheelchair Session
Number analyzed (Participants) | 14 | 9 | 11 | 11
scores on a scale
  Q1. (session1) 1: A lot, 5: A little | 2.57 (1.16) | 2.78 (0.67) | 2.91 (1.38) | 3.10 (1.29)
  Q1. (session2) 1: A lot, 5: A little | 4.07 (0.83) | 3.44 (1.13) | 3.90 (1.10) | 3.91 (0.70)
  Q1. (session3) 1: A lot, 5: A little | 4.25 (0.87) | 3.56 (1.01) | 3.82 (0.87) | 4.00 (1.10)
  Q1. (session4) 1: A lot, 5: A little | 4.50 (0.80) | 3.63 (1.06) | 3.91 (1.30) | 3.73 (1.35)
  Q1. (session5) 1: A lot, 5: A little | 4.17 (0.96) | 3.33 (1.00) | 4.27 (0.90) | 4.09 (1.83)
  Q1. (session6) 1: A lot, 5: A little | NA (NA) — Group-A subjects completed 5-session trials. | NA (NA) — Group-B subjects completed 5-session trials. | 4.36 (0.81) | NA (NA) — Group-C subjects were asked about wheelchair related questionnaire only for 5-session trials.
  Q2. (session1) 1: Too slow, 3: Just right, 5: Too | 3.21 (0.43) | 3.11 (0.78) | 3.27 (0.47) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q2. (session2) 1: Too slow, 3: Just right, 5: Too | 3.07 (0.47) | 3.22 (1.09) | 0.34 (0.52) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q2. (session3) 1: Too slow, 3: Just right, 5: Too | 3.00 (0.43) | 3.22 (1.30) | 3.00 (0.89) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q2. (session4) 1: Too slow, 3: Just right, 5: Too | 3.00 (0.43) | 3.13 (0.64) | 3.27 (0.79) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q2. (session5) 1: Too slow, 3: Just right, 5: Too | 3.08 (0.49) | 3.00 (0.71) | 3.18 (0.75) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q2. (session6) 1: Too slow, 3: Just right, 5: Too | NA (NA) — Group-A subjects completed 5-session trials. | NA (NA) — Group-B subjects completed 5-session trials. | 3.18 (0.75) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q3. (session1) 1: Very difficult, 5: Very easy | 2.71 (0.73) | 3.56 (0.88) | 3.36 (1.12) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q3. (session2) 1: Very difficult, 5: Very easy | 3.43 (0.94) | 2.89 (0.60) | 3.90 (0.57) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q3. (session3) 1: Very difficult, 5: Very easy | 3.50 (0.80) | 3.11 (0.78) | 3.64 (0.81) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q3. (session4) 1: Very difficult, 5: Very easy | 3.92 (0.67) | 3.75 (0.71) | 3.91 (0.70) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q3. (session5) 1: Very difficult, 5: Very easy | 4.15 (0.69) | 3.00 (0.71) | 4.09 (0.83) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q3. (session6) 1: Very difficult, 5: Very easy | NA (NA) — Group-A subjects completed 5-session trials. | NA (NA) — Group-B subjects completed 5-session trials. | 4.27 (0.79) | NA (NA) — This questionnaire does not contain the computer related questions.
  Q4.(ses1)1:Very difficult,5:Very easy(GrpC:Q4-1) | 3.43 (0.76) | 3.22 (1.20) | NA (NA) — This questionnaire does not contain the PWC related questions. | 4.10 (0.88)
  Q4.(ses2)1:Very difficult,5:Very easy(GrpC:Q4-1) | 3.93 (0.62) | 4.11 (0.78) | NA (NA) — This questionnaire does not contain the PWC related questions. | 4.00 (0.77)
  Q4.(ses3)1:Very difficult,5:Very easy(GrpC:Q4-1) | 3.75 (0.87) | 3.44 (0.88) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.64 (1.12)
  Q4.(ses4)1:Very difficult,5:Very easy(GrpC:Q4-1) | 4.25 (0.97) | 3.50 (1.69) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.73 (1.01)
  Q4.(ses5)1:Very difficult,5:Very easy(GrpC:Q4-1) | 4.07 (0.92) | 3.67 (1.12) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.82 (0.75)
  Q5. (session1) 1: Too slow, 5: Too Fast | 2.71 (0.47) | 2.67 (0.87) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.70 (0.67)
  Q5. (session2) 1: Too slow, 5: Too Fast | 2.29 (0.61) | 2.44 (0.73) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.64 (0.92)
  Q5. (session3) 1: Too slow, 5: Too Fast | 2.58 (0.67) | 2.22 (0.67) | NA (NA) — This questionnaire does not contain the PWC related questions. | 0.64 (0.81)
  Q5. (session4) 1: Too slow, 5: Too Fast | 2.50 (0.67) | 2.25 (0.46) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.55 (0.82)
  Q5. (session5) 1: Too slow, 5: Too Fast | 2.36 (0.63) | 1.78 (0.67) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.27 (1.01)
  Q6. (session1) 1: Very jerky, 5: Very smooth | 4.14 (0.77) | 3.67 (1.12) | NA (NA) — This questionnaire does not contain the PWC related questions. | 4.00 (0.94)
  Q6. (session2) 1: Very jerky, 5: Very smooth | 4.14 (0.86) | 3.33 (0.71) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.91 (1.14)
  Q6. (session3) 1: Very jerky, 5: Very smooth | 4.50 (0.80) | 3.22 (0.97) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.91 (1.04)
  Q6. (session4) 1: Very jerky, 5: Very smooth | 4.08 (1.08) | 3.63 (0.92) | NA (NA) — This questionnaire does not contain the PWC related questions. | 4.00 (1.10)
  Q6. (session5) 1: Very jerky, 5: Very smooth | 4.00 (1.11) | 3.63 (0.92) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.82 (1.08)
  Q4.(ses1)1:Very difficult,5:Very easy(GrpC:Q4-2) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.20 (0.79)
  Q4.(ses2)1:Very difficult,5:Very easy(GrpC:Q4-2) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.45 (1.13)
  Q4.(ses3)1:Very difficult,5:Very easy(GrpC:Q4-2) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.91 (0.70)
  Q4.(ses4)1:Very difficult,5:Very easy(GrpC:Q4-2) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.64 (1.36)
  Q4.(ses5)1:Very difficult,5:Very easy(GrpC:Q4-2) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.91 (0.83)
  Q4.(ses1)1:Very difficult,5:Very easy(GrpC:Q4-3) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.40 (1.43)
  Q4.(ses2)1:Very difficult,5:Very easy(GrpC:Q4-3) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.73 (1.27)
  Q4.(ses3)1:Very difficult,5:Very easy(GrpC:Q4-3) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 4.00 (0.89)
  Q4.(ses4)1:Very difficult,5:Very easy(GrpC:Q4-3) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 4.00 (1.00)
  Q4.(ses5)1:Very difficult,5:Very easy(GrpC:Q4-3) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 3.64 (0.92)
  Q4.(ses1)1:Very difficult,5:Very easy(GrpC:Q4-4) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.70 (0.67)
  Q4.(ses2)1:Very difficult,5:Very easy(GrpC:Q4-4) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.64 (0.92)
  Q4.(ses3)1:Very difficult,5:Very easy(GrpC:Q4-4) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.64 (0.81)
  Q4.(ses4)1:Very difficult,5:Very easy(GrpC:Q4-4) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.55 (0.82)
  Q4.(ses5)1:Very difficult,5:Very easy(GrpC:Q4-4) | NA (NA) — This question was not separately asked for Group-A PWC session. (Check Q4) | NA (NA) — This question was not separately asked for Group-B PWC session. (Check Q4) | NA (NA) — This questionnaire does not contain the PWC related questions. | 2.27 (1.01)
  Q7.(ses1)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have phone dialing task. | NA (NA) — Group-B subjects did not have phone dialing task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 3.22 (1.86)
  Q7.(ses2)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have phone dialing task. | NA (NA) — Group-B subjects did not have phone dialing task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 4.00 (1.41)
  Q7.(ses3)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have phone dialing task. | NA (NA) — Group-B subjects did not have phone dialing task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 4.10 (1.37)
  Q7.(ses4)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have phone dialing task. | NA (NA) — Group-B subjects did not have phone dialing task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 4.40 (1.07)
  Q7.(ses5)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have phone dialing task. | NA (NA) — Group-B subjects did not have phone dialing task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 4.80 (0.63)
  Q8.(ses1)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have weight shifting task. | NA (NA) — Group-B subjects did not have weight shifting task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 3.71 (1.70)
  Q8.(ses2)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have weight shifting task. | NA (NA) — Group-B subjects did not have weight shifting task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 4.60 (0.97)
  Q8.(ses3)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have weight shifting task. | NA (NA) — Group-B subjects did not have weight shifting task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 4.70 (0.67)
  Q8.(ses4)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have weight shifting task. | NA (NA) — Group-B subjects did not have weight shifting task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 4.70 (0.67)
  Q8.(ses5)1:Completely ineffective,5:Very effective | NA (NA) — Group-A subjects did not have weight shifting task. | NA (NA) — Group-B subjects did not have weight shifting task. | NA (NA) — This questionnaire does not contain the smartphone related questions. | 4.70 (0.67)

ADVERSE EVENTS:
Arm/Group | Able-bodied Subject With Tongue Piercing (Group-A) | Able-bodied Subject Without Tongue Piercing (Group-B) | Subjects With Spinal Cord Injury (Group-C)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/16 | 0/24 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No